CLINICAL TRIAL: NCT04160247
Title: Clinical Evaluation of Cemented and Angulated Screw-retained Crowns Following Immediate Implant Placement: a Randomized Controlled Clinical Trials
Brief Title: Angulated Screw-retained Crowns Following Immediate Implant Placement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH9-19-07
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Tooth Diseases
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angulated screw-retained crown (Active Comparator): Restorations are connected to the implants by angulated screw channel system
  Interventions: Procedure: Immediate implant placement; Procedure: Angulated screw-retained crowns placement
- Cemented crown (Placebo Comparator): Restorations are cemented onto the implant abutment
  Interventions: Procedure: Immediate implant placement; Procedure: Cemented crowns placement

INTERVENTIONS:
Procedure: Immediate implant placement — Implants are placed in fresh socket
Procedure: Angulated screw-retained crowns placement — To insert the restorations by angulated screw systems
  Arms: Angulated screw-retained crown
Procedure: Cemented crowns placement — To cement the restorations onto the implant abutment
  Arms: Cemented crown

SUMMARY:
There are two choices of restorations and implant abutments connection now: cemented and screw-retained.The excess cement, which would be difficult to completely remove, might lead to series of biological complications. The angulated screw channel (ASC) abutments, which recently introduced by Nobel Biocare , largely address the problem with visible screw access that may compromise esthetics. However, all of the present studies were clinical reports, thus the clinical efficacy of ASC abutments still needs the verification of evidence-based medicine with larger sample. Therefore, we designed a randomized controlled clinical trial study, aiming to verify the clinical efficacy of the ASC abutments by comparing screw-retained (with ASC abutments) single implant crowns with cemented ones in esthetic region.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and in good health;
2. Single tooth implant (type 1) in the esthetic region;
3. Patients with natural teeth adjacent to single implant crowns;
4. Patients with periodontal treatment before implant surgery;
5. The implants are from Nobel Biocare system with tapered link and the permanent restoration is a single crown and all-ceramic;
6. Soft tissue in the implanting-and-adjacent areas is healthy and free of infection

Exclusion Criteria:

1. Multiple implants in the esthetic region, or the restoration is a bridge
2. Patients with bone augmentation procedures;
3. Heavy smokers (>10 cigarettes/day);
4. Medically compromised patients (American Society of Anesthesiologists (ASA) classification III-IV);
5. Implants in an incorrect three-dimensional position (definition according to ITI VOL1);
6. Uncontrolled diabetes mellitus;
7. Unwilling to participate in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
BOP% | from baseline to 1-year follow-up
  Percentage of bleeding on probing positive

SECONDARY OUTCOMES:
PPD | from baseline to 1-year follow-up
  Pocket probing depth
MBL | from baseline to 1-year follow-up
  Marginal bone loss
PES | from baseline to 1-year follow-up
  pink esthetic score

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai NinthPeoples' Hospital, Shanghai, China